CLINICAL TRIAL: NCT05839587
Title: Short-term Outcome and Inflammatory Stress Response Following Transabdominal Preperitoneal Inguinal Hernia Repair (TAPP) - A Prospective, Randomized Trial Comparing Laparoscopy to the Robotic-assisted Approach
Brief Title: Transabdominal Preperitoneal Inguinal Hernia Repair
Acronym: TAPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS-MT Kir - 1 - 2023
Record Dates: First submitted 2023-02-28; First posted 2023-05-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Hernia, Inguinal; Laparoscopy
Keywords: Adult; Robotic surgical procedures; Abdomen
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic TAPP (Experimental): Repair of primary unilateral and bilateral hernias with robotic technology
  Interventions: Procedure: Robotic TAPP
- Laparoscopic TAPP (Active Comparator): Repair of primary unilateral and bilateral hernias with laparoscopic repair
  Interventions: Procedure: Laparoscopic TAPP

INTERVENTIONS:
Procedure: Robotic TAPP — Robotic TAPP consists of four different procedures. Part 2 and 3 will be the same for both procedures and will consist of hernia reduction and preparation of the preperitoneal space where the mesh is placed (part 2), mesh placement and suturing of the peritoneum (part 3). Part 1 consists of docking of the robot and port placement and part 4 consists of de-docking and skin closure
  Arms: Robotic TAPP
Procedure: Laparoscopic TAPP — Laparoscopic TAPP consists of four different procedures. Part 2 and 3 will be the same for both procedures and will consist of hernia reduction and preparation of the preperitoneal space where the mesh is placed (part 2), mesh placement and suturing of the peritoneum (part 3). Part 1 consists of port placement only and part 4 consists of skin closure only.
  Arms: Laparoscopic TAPP

SUMMARY:
The present study seeks to determine whether improved visual acuity and enhanced flexibility of the robotic platform results in a reduced surgical stress response and an improvement in indices of surgical outcome measures for simple and complex inguinal hernia repair

DETAILED DESCRIPTION:
Complex inguinal hernia repair is challenging and requires both advanced skills in laparoscopic surgery and knowledge about the complex anatomy of the inguinal area. Whereas the repair of a small inguinal hernia usually is simple and straightforward, complex hernias (large inguinoscrotal and recurrent hernias) constitute a surgical challenge due to the risk of damage of the neurovascular structures in the inguinal area. It requires advanced laparoscopic skills to reduce the hernial sac in patients with large lateral hernias, where the hernial sac often extends deep into the scrotum in close vicinity to the spermatic cord and the testicular artery. This dissection is difficult with conventional laparoscopy, which may explain the risk of chronic pain, testicular hypotrophy and hernia recurrence. The aim of the study is to determine whether rTAPP of complex inguinal hernias is associated with a lower surgical stress response and a lower risk of postoperative complications compared to laparoscopic TAPP.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1- 3
* Clinical or radiologic diagnosis of inguinal hernia (unilateral, bilateral, recurrent, inguinoscrotal)
* Eligible for a laparoscopic procedure
* Informed concent

Exclusion Criteria:

* Incarcerated inguinal hernia requiring emergency surgery
* Pregnancy
* Patients with chronic pain due to arthritis, migraine or other illness requiring regular intake of pain relieve (paracetamol, NSAID etc)
* Active cancer
* History of psychiatric or additive disorder that prevent the patient from participating in the trial
* Co-existing inflammatory disease
* Co-existing immunological disease that requires medication of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Surgical stress response (CRP) | CRP will be measured preoperatively at baseline, 1 day postoperatively and 3 days postoperatively
  Change of serum CRP over time.

SECONDARY OUTCOMES:
Estimated intraoperative blood loss | intraoperative (From first incision until last suture has been placed)
  The amount of intraoperative blood loss measured in mL, estimated by the primary surgeon
Intraoperative need of blood transfusion | intraoperative (From first incision until last suture has been placed)
  The amount of blood transfused during surgery measured in mL
Length of hospital stay | Up to 3 months
  The number of days patients spend in the hospital following the procedure.
Hernia defect size | During surgery
  The area of the hernial defect in cm2 measured at 8 mmHg
Total surgical time | During surgery
  The procedure will be divided into 4 parts. Part 1 will be different for the 2 procedures. In rTAPP it will consist of docking of the robot and port placement while it only will consist of port placement in TAPP. Part 2 and 3 will be the same for both procedures and will consist of hernia reduction and preparation of the preperitoneal space where the mesh is placed (part 2), mesh placement and suturing of the peritoneum (part 3). Part 4 will also be different for the 2 procedures. In rTAPP it will consist of de-docking and skin closure while it only will consist of skin closure in TAPP. Total surgical time and each part will be measured individually in minutes and the 2 procedures will be compared
Postoperative complications | From surgery until 6 months postoperatively
  Classified into grades (I-V) according to the Clavien-Dindo classification
Life-quality | From inclusion until 6 months postoperatively
  According to the EUropean Registry for Abdominal wall HerniaS Quality Of Life questionnaire (Eura-HS QoL). The total score ranges from 0 (best quality of life) to 90 (worst quality of life)
Sexual dysfunction | From inclusion until 6 months postoperatively
  According to the Sexual Inguinal Hernia Questionnaire (SexIHQ) a 1-page, 8-question questionnaire including visual analogue scales and tick-boxes used to asses sexual dysfunction following inguinal hernia repair
Surgical stress response (IL1-β) | IL1-β will be measured preoperatively at baseline, 30 minutes after extubation and 120 minutes after extubation
  The change of serum IL1-β over time.
Surgical stress response (IL-6) | IL-6 will be measured preoperatively at baseline, 30 minutes after extubation and 120 minutes after extubation
  The change of serum IL-6 over time.
Surgical stress response (IL-8) | IL-8 will be measured preoperatively at baseline, 30 minutes after extubation and 120 minutes after extubation
  The change of serum IL-8 over time.
Surgical stress response (IL-10) | IL-10 will be measured preoperatively at baseline, 30 minutes after extubation and 120 minutes after extubation
  The change of serum IL-10 over time.
Surgical stress response (TNF-α) | TNF-α will be measured preoperatively at baseline, 30 minutes after extubation and 120 minutes after extubation
  The change of serum TNF-α over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCormack K, Scott NW, Go PM, Ross S, Grant AM; EU Hernia Trialists Collaboration. Laparoscopic techniques versus open techniques for inguinal hernia repair. Cochrane Database Syst Rev. 2003;2003(1):CD001785. doi: 10.1002/14651858.CD001785. PMID 12535413
- [Background] Podolsky D, Novitsky Y. Robotic Inguinal Hernia Repair. Surg Clin North Am. 2020 Apr;100(2):409-415. doi: 10.1016/j.suc.2019.12.010. Epub 2020 Feb 1. PMID 32169186
- [Background] Huerta S, Timmerman C, Argo M, Favela J, Pham T, Kukreja S, Yan J, Zhu H. Open, Laparoscopic, and Robotic Inguinal Hernia Repair: Outcomes and Predictors of Complications. J Surg Res. 2019 Sep;241:119-127. doi: 10.1016/j.jss.2019.03.046. Epub 2019 Apr 22. PMID 31022677
- [Derived] Valorenzos A, Nielsen KA, Kaiser K, Petersen SR, Helligso P, Dorfelt A, Lambertsen KL, Ellebaek MB, Nielsen MF. Inflammatory response and short-term outcomes after laparoscopic versus robotic transabdominal preperitoneal inguinal hernia repair: randomized clinical trial (ROLAIS). Br J Surg. 2025 Mar 28;112(4):znaf074. doi: 10.1093/bjs/znaf074. PMID 40277023
- [Derived] Valorenzos AV, Nielsen KA, Kaiser K, Helligso P, Ellebaek MB, Dorfelt A, Petersen SR, Pedersen AK, Nielsen MF. Short-term outcomes and inflammatory stress response following laparoscopy or robotic-assisted transabdominal preperitoneal inguinal hernia repair (TAPP): study protocol for a prospective, randomized trial (ROLAIS). Trials. 2024 Aug 8;25(1):529. doi: 10.1186/s13063-024-08361-w. PMID 39118135